CLINICAL TRIAL: NCT00430729
Title: Effect of Roflumilast on Exacerbation Rate in Patients With Chronic Obstructive Pulmonary Disease. A 52 Weeks Double Blind Study With 500mcg Roflumilast Once Daily Versus Placebo. Ratio-Study.
Brief Title: Effect of Roflumilast on Exacerbation Rate in Patients With Chronic Obstructive Pulmonary Disease. Ratio-Study. (BY217/M2-112)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BY217/M2-112
Record Dates: First submitted 2007-02-01; First posted 2007-02-02 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Obstructive Pulmonary Disease; COPD
Keywords: Roflumilast
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Roflumilast

INTERVENTIONS:
Drug: Roflumilast

SUMMARY:
The purpose of this study is to investigate the effect of 500mcg roflumilast vs placebo on exacerbation rate and pulmonary function as well as quality of life in patients with chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Main Inclusion Criteria:

* FEV1/FVC ratio (post-bronchodilator) ≤70%
* FEV1 (post-bronchodilator) ≤50% of predicted
* Current smoker or ex-smoker
* Clinically stable COPD indicated by no exacerbation and no change in COPD treatment of within 4 weeks prior to baseline
* Availability of a chest x-ray dated a maximum of 6 months prior to study baseline visit B0 or a willingness to have a chest x-ray performed before baseline

Main Exclusion Criteria:

* COPD exacerbation indicated by a treatment with systemic glucocorticoids not stopped 4 weeks prior to baseline
* Lower respiratory tract infection not resolved 4 weeks prior to baseline
* Diagnosis of asthma and/or other relevant lung disease
* Known alpha-1-antitrypsin deficiency
* Need for long-term oxygen therapy defined as ≥16 hours/day

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100
Dates: Start 2003-01

PRIMARY OUTCOMES:
The frequency of patients experiencing at least one moderate or severe exacerbation during the treatment period.
Change in FEV1 from baseline during the treatment period.

SECONDARY OUTCOMES:
Pulmonary function variables; quality of life variables;patient diary variables;safety

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (14):
- ALTANA Pharma, Cities in Australia, Australia
- ALTANA Pharma, Cities in Austria, Austria
- ALTANA Pharma, Cities in Canada, Canada
- ALTANA Pharma, Cities in France, France
- ALTANA Pharma, Cities in Hungary, Hungary
- ALTANA Pharma, Cities in Italy, Italy
- ALTANA Pharma, Cities in the Netherlands, Netherlands
- ALTANA Pharma, Cities in Poland, Poland
- ALTANA Pharma, Cities in Portugal, Portugal
- ALTANA Pharma, Cities in the Russian Federation, Russia
- ALTANA Pharma, Cities in South Africa, South Africa
- ALTANA Pharma, Cities in Spain, Spain
- ALTANA Pharma, Cities in Switzerland, Switzerland
- ALTANA Pharma, Cities in the United Kingdom, United Kingdom

REFERENCES:
- [Derived] Facius A, Krause A, Claret L, Bruno R, Lahu G. Modeling and Simulation of Pivotal Clinical Trials Using Linked Models for Multiple Endpoints in Chronic Obstructive Pulmonary Disease With Roflumilast. J Clin Pharmacol. 2017 Aug;57(8):1042-1052. doi: 10.1002/jcph.885. Epub 2017 Apr 17. PMID 28419462
- [Derived] Rennard SI, Calverley PM, Goehring UM, Bredenbroker D, Martinez FJ. Reduction of exacerbations by the PDE4 inhibitor roflumilast--the importance of defining different subsets of patients with COPD. Respir Res. 2011 Jan 27;12(1):18. doi: 10.1186/1465-9921-12-18. PMID 21272339
- See also: BY217-M2-112-RDS-2005-05-11.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4478&filename=BY217-M2-112-RDS-2005-05-11.pdf